CLINICAL TRIAL: NCT01515540
Title: Brain Imaging of Lidoderm for Chronic Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU00022968
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Low Back Pain
Keywords: chronic back pain; placebo; fmri; brain imaging
MeSH Terms: conditions — Low Back Pain | interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine (Active Comparator): 5% lidoderm patch
  Interventions: Drug: lidocaine
- control (Placebo Comparator): placebo patch
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lidocaine — 5% lidoderm patch
  Other Names: Lidoderm (Endo Pharmaceuticals); 5% lidocaine patch
  Arms: lidocaine
Drug: placebo — placebo
  Other Names: sham patch
  Arms: control

SUMMARY:
The investigators tested whether pain decrease can be observed centrally with non-invasive brain imaging in CBP subjects receiving Lidoderm. The investigators first tested effects of 5% Lidoderm patched in an open labelled trial. Next the investigators compared the effects of Lidocaine versus Placebo patches. Three time points were evaluated: baseline (before treatment) and 6 hours and 2 weeks after treatment. The latter trial was a 2 arm, double blind, placebo controlled trial, where participants either received Lidoderm or placebo patches, without cross over.

DETAILED DESCRIPTION:
Previous data showed that Lidoderm patches that contain 5% Lidocaine applied to the affected area for a period of 1-2 weeks decreased chronic pain. We conducted a preliminary open-label trial in chronic back pain patients and found that the patients reported reduction in pain intensity and associated brain activity (measured with fMRI). As a next step, we conducted a double blind clinical trial where the drug was tested against placebo to determine whether the effects on CBP were mediated by a pharmacological mechanism. For this we obtained psychophysical measurements of pain and measures of brain activity using fMRI. Two scans after treatment (6 hour and 2 weeks after treatment) were conducted to observe the effects of short term and long term use.

Brain activity was measured by the non-invasive method of functional imaging (fMRI), which enables examination of cortical blood flow during pain rating. These brain scans were acquired in chronic back pain patients while they rated their ongoing chronic pain using a finger span device. In a control task, each patient also rated the changes in the length of a bar n a screen (a visual control task). Anatomical scans were also acquired.

The general design of the study was that CBP subjects were assesses with fmri for brain responses for ongoing pain at three time points. The initial (baseline) scan occurred after a minimum of 48 hour period during which the patients refrained from taking analgesic medication. The patients were next scanned at 6 hours after treatment and again after 2 weeks of continuous treatment. Subjects were randomised to placebo or Lidoderm (both Lidoderm and placebo patches were supplied by Endo Pharmaceuticals).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 18 years or older of age
2. Pain in the location of the lower back
3. Pain duration for a minimum of 6 months on a continuous basis
4. Pain intensity of at least 3 out of 10 on most days of the week over the past six months
5. Manifestations of radicular element of pain: radiation below knee (examples towards thigh, buttocks).
6. Right handedness

Exclusion Criteria:

1. Applying for or currently receiving workers' compensation or disability status.
2. Back pain secondary to spinal cord injury
3. Back pain secondary to any systemic condition (e.g ankylosing spondylitis0
4. Diabetes mellitus
5. Back pain secondary to tumors.
6. Standard MRI criteria re: claustrophobia, metal objects etc.
7. Subjects with cognitive deficits such as dementia, psychiatric illness including depression with a BDI score of more than 19 (moderate to severe depression), history of brain injury, history of chronic disease
8. Pregnant and/or lactating women
9. Left handedness
10. Active cancer
11. Other serious painful condition (e.g., arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apkar V. Apkarian, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Baliki MN, Geha PY, Jabakhanji R, Harden N, Schnitzer TJ, Apkarian AV. A preliminary fMRI study of analgesic treatment in chronic back pain and knee osteoarthritis. Mol Pain. 2008 Oct 25;4:47. doi: 10.1186/1744-8069-4-47. PMID 18950528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients were recruited for the brain imaging and treatment study. Data from 7 subjects was not analyzed due to failure to attend the repeat sessions for non specific reasons and data from 1 subject was excluded from analysis due to technical faults. Thus, data from a total of 30 subjects was included in the brain imaging analysis.
Period: Overall Study
Arm/Group | Lidocaine | Control
Started | 20 | 18
Completed | 15 | 15
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Control | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (7.7) | 49.73 (10.27) | 51.36 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity on a Visual Analog Scale (VAS) The Scale Had Values From 0-100, Where 0 Represents "no Pain" and 100 Was the "Worst Pain Imaginable".
Description: the primary hypothesis was that the lidoderm 5% patch was expected to decrease pain intensity post treatment greater than placebo patch.
  A lower value on the 0-100 scale is considered to represent less pain. Higher values represent more pain. Greater than 20%-30% decrease in pain is considered clinically meaningful.
Time Frame: 2 weeks
Population: based on a literature search.
Measure: Mean (Standard Deviation); unit: peak pain intensity
Arm/Group | Lidocaine | Control
Number analyzed (Participants) | 15 | 15
peak pain intensity | 51.0 (7.6) | 51.6 (7.1)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Lidocaine | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No